CLINICAL TRIAL: NCT02602678
Title: Prone Position Effects on Work of Breathing and Intrinsic PEEP in Children With Severe Acute Viral Bronchiolitis
Acronym: BRONCHIO-DV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL15_0430
Record Dates: First submitted 2015-11-09; First posted 2015-11-11 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Severe Bronchiolitis
Keywords: Children.; prone position; acute viral bronchiolitis; syncytial virus; work of breathing; intrinsic PEEP
MeSH Terms: conditions — Bronchiolitis; Positive-Pressure Respiration, Intrinsic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRONE-Supine (Experimental): We test the hypothesis that in infants with severe bronchiolitis, prone position reduces the work of breathing (WOB) and the intrinsic Positive End Expiratory Pressure (PEEP).
  Interventions: Procedure: Prone then supine position
- SUPINE - Prone (Experimental): We test the hypothesis that in infants with severe bronchiolitis, prone position reduces the work of breathing (WOB) and the intrinsic Positive End Expiratory Pressure (PEEP).
  Interventions: Procedure: Supine then Prone position

INTERVENTIONS:
Procedure: Supine then Prone position — One hour in supine position with CPAP (+7 cmH2O) then 15 min in supine position in spontaneous ventilation (wash-out) and one hour in prone position with CPAP (+7 cmH2O)
  Arms: SUPINE - Prone
Procedure: Prone then supine position — One hour in prone position with CPAP (+7 cmH2O) then 15 min in supine position in spontaneous ventilation (wash out ) and one hour in supine position with CPAP (+7 cmH2O)
  Arms: PRONE-Supine

SUMMARY:
Acute viral bronchiolitis is the first cause of respiratory distress in infant. Airway inflammation increases the respiratory system resistances and dynamic hyperinflation. This leads to an increase in the work of breathing. In Chronic obstructive pulmonary disease patients as in neonates, prone position (PP) improves lung function and decreases the end expiratory lung volume. The investigators hypothesized that in infants with severe bronchiolitis, prone position reduces the intrinsic Positive End Expiratory Pressure (PEEPi) and the work of breathing (WOB). The investigator designed a prospective randomized crossover study with 16 infants younger than six months who need ventilatory support by nasal continuous positive airway pressure (nCPAP) for severe acute viral bronchiolitis. Work of breathing (product time pressure) and PEEPi will be estimated using an esophageal pressure probe in prone and supine position.

ELIGIBILITY:
Inclusion Criteria:

* Infant < 6 months
* Admitted in the pediatric intensive care unit of the Femme-Mère-Enfant hospital, Hospices Civils de Lyon, France
* With severe acute viral bronchiolitis requiring ventilatory support (mWCAS > 4 and/or and or FiO2> 40% and/or hypercapnic acidosis (pH<7.30 and/or pCO2>8 kPa))
* Signed informed consent by the two parents or the owner of parental authority

Exclusion Criteria:

* Chronic respiratory, neuromuscular, ENT or cardiac disease
* Contraindication for placement of esophageal probe (esophageal surgery, varices, …)
* Children requiring invasive ventilation (more than 3 significant apneas in 1 hour, decreased consciousness, …)
* Children not affiliated to a social security scheme

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2015-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Work of breathing | 60 min
  The primary outcome is the work of breathing (WOB) estimated by the mean on 100 breaths of the esophageal and trans-diaphragmatic Pressure-Time Product (PTP) at the end of the first hour.

SECONDARY OUTCOMES:
Intrinsic PEEP | 60 min
  Mean on 10 breaths of the intrinsic positive end expiratory pressure in spontaneous ventilation
Inspiratory:Expiratory Time Ratio | 60 min
  Mean on 100 breaths of the Inspiratory:Expiratory Time Ratio
Heart rate | 60 min
  Evolution of the clinical and oxygenation parameter within the first hour in each position.
Respiratory rate | 60 min
  Evolution of the clinical and oxygenation parameters within the first hour in each position.
SPO2 | 60 min
  Evolution of the clinical and oxygenation parameters within the first hour in each position.
Transcutaneous CO2 | 60 min
  Evolution of the clinical and oxygenation parameters within the first hour in each position.
EDIN score (neonatal pain and discomfort scale) | 60 min

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Bron, France

REFERENCES:
- [Result] Baudin F, Emeriaud G, Essouri S, Beck J, Portefaix A, Javouhey E, Guerin C. Physiological Effect of Prone Position in Children with Severe Bronchiolitis: A Randomized Cross-Over Study (BRONCHIO-DV). J Pediatr. 2019 Feb;205:112-119.e4. doi: 10.1016/j.jpeds.2018.09.066. Epub 2018 Nov 14. PMID 30448014